CLINICAL TRIAL: NCT00293293
Title: Outcomes in Ovarian Cancer and Fallopian Tube Cancer Patients Using Complementary Alternative Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Randy Shaver Cancer Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000NT790; UMN-WCC-30 (Other: Women's Cancer Center, University of Minnesota); 0012M77821 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Results first posted 2012-06-06 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer; Peritoneal Primary Cancer; Fallopian Tube Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Touch; Massage; Hypnosis; Mind-Body Therapies; taxane; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy Alone (Active Comparator): Patients receiving 6 cycles of taxane and platinum therapy for ovarian, fallopian tube or primary peritoneal cancer by their treating physician. Chemotherapy administration is not administered as part of this protocol.
  Interventions: Drug: Standard chemotherapy
- Standard Chemotherapy + CAM (Experimental): Patients receiving 6 cycles of taxane and platinum therapy for ovarian, fallopian tube or peritoneal cancer with additional complementary alternative medicine - CAM (healing touch, hypnosis and massage therapy). Chemotherapy administration is not administered as part of this protocol.
  Interventions: Other: healing touch; Other: massage therapy; Other: hypnosis

INTERVENTIONS:
Other: healing touch — The practitioner performed a structured interview with the patient both a verbal assessment and an energy/physical assessment using pendulum and hand scan techniques. The practitioner will then provide the intervention which will consist of: chakra connection, magnetic passes (hands still and in motion), magnetic clearing.
  Other Names: energy-based therapy
  Arms: Standard Chemotherapy + CAM
Other: massage therapy — Standard massage techniques will be employed over the head, neck, shoulders, back, hands, and/or feet areas. The intensity and rapidity of massage movements will be individualized to the patient's comfort level.
  Other Names: massage
  Arms: Standard Chemotherapy + CAM
Other: hypnosis — Steps: 1) begins with a progressive relaxation induction; 2) suggestions for deepening are then provided; 3) offered suggestions to increase comfort with medical procedures; 4) suggestion for enhanced capacity for coping will be given as an ego strengthening suggestion, with a post-hypnotic suggestion for increasing comfort/success in coping each time.
  Other Names: mind-body intervention procedure
  Arms: Standard Chemotherapy + CAM
Drug: Standard chemotherapy — Patients will receive 6 cycles of taxane and platinum therapy as prescribed by their treating physician. Chemotherapy treatment is not part of this study.
  Other Names: Taxane; Platinum
  Arms: Chemotherapy Alone

SUMMARY:
RATIONALE: Chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hypnosis, massage therapy, and healing touch may improve the quality of life of patients who are undergoing chemotherapy.

PURPOSE: This randomized clinical trial is studying how well giving hypnosis, massage therapy and healing touch changes outcomes in women receiving chemotherapy for newly diagnosed epithelial ovarian, fallopian tube or peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether quality of life is improved in patients with epithelial ovarian, fallopian tube or primary peritoneal cavity cancer receiving hypnosis, massage therapy, and healing touch and standard chemotherapy as compared to patients receiving standard chemotherapy alone.

Secondary

* Determine changes in immunologic response markers, chemotherapy side effects, and complication rates in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard therapy): Patients undergo standard chemotherapy for epithelial ovarian, fallopian tube or primary peritoneal cancer.
* Arm II (standard therapy with complementary alternative medicine): Patients undergo chemotherapy as in arm I. Patients also undergo massage over approximately 30 minutes and healing touch therapy over approximately 30 minutes with each course of chemotherapy 1-6 and hypnosis over 30-60 minutes during courses 1, 2, and 4.

Quality of life is assessed at baseline, during courses 3 and 6 of chemotherapy, and then 6 months after completion of study treatment.

After completion of study treatment, patients are followed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed epithelial ovarian, primary peritoneal or fallopian tube cancer, any pathologic type or stage, who will receive 6 cycles of chemotherapy.
* Patients must have signed an informed consent

Exclusion Criteria:

* Previous cancer other than skin cancer
* Previous chemotherapy experience
* Active substance abuse
* Schizophrenia
* Pregnant or lactating

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-05; Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Judson, MD, Study Chair — Moffitt
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients made informed consent and were randomized to chemotherapy alone or chemotherapy with complementary alternative medicine (hypnosis, massage, healing touch). Patients received either intravenous paclitaxel and carboplatin on an every 3 week basis, or a combination of intravenous and intraperitoneal paclitaxel and cisplatin.
Pre-assignment Details: Analysis was conducted as intent-to-treat. All randomized patients were included, regardless of number of courses of chemotherapy, CAM therapy or survival. All women in the CAM arm of the trial received all prescribed CAM interventions. No investigational drugs were administered as a part of this protocol.
Groups:
- Chemotherapy Alone: Patients receiving 6 cycles of a taxane or platinum therapy for ovarian, peritoneal, or fallopian tube cancer by their treating physician.
- Chemotherapy + CAM: Patients receiving 6 cycles of a taxane or platinum therapy therapy for ovarian, peritoneal, or fallopian tube cancer with additional complementary alternative medicine - CAM (hypnosis, healing touch and massage therapy).
Period: Overall Study
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Started | 20 | 23
Completed | 18 | 21
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Patient "too anxious" to complete trial | 1 | 0
Not completed — Patient discontinued chemotherapy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 27
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (11.4) | 58.8 (11.8) | 60.72 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Comparison - Average FACT-O Scoring in Chemotherapy Alone vs. Chemotherapy Plus Complementary Alternative Medicine (CAM)
Description: Measured by Functional Assessment of Cancer Therapy-Ovarian (FACT-O) questionnaire was used to assess patients' quality of life before each chemotherapy cycle. It is a standardized self-administered questionnaire measuring many aspects of quality of life (0 to 4; Not at all, A little bit, Some-what, Quite a bit, Very much) as related to patients with ovarian cancers. The quality of life measures include the total FACT-O score (minimum value 0, maximum value 200). Questionnaires are recoded in the final analysis phase so that a higher score reflected more adverse effects on quality of life.
Time Frame: Prior to Cycle 1 (Day -2 to +1), Every 3rd cycle (1 cycle = approx 21 days) and 6 Months Post Chemotherapy
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
Scores on a Scale
  Prior to Cycle 1 | 143 [121 to 200] | 152 [138 to 187]
  Prior to Cycle 3 | 154 [120 to 179] | 152 [101 to 184]
  Prior to Cycle 6 | 158 [141 to 188] | 152 [119 to 200]
  6 Months Post Chemotherapy (+/- 15 days) | 173 [98 to 190] | 162 [155 to 200]

2. Primary Outcome: Comparison of Mental Health Inventory (MHI) Questionnaire Results - Average for Chemotherapy Alone vs. Chemotherapy Plus CAM
Description: The MHI asks questions about how the consumer is feeling and coping with usual life activities. It provides measurable information about the consumer's wellbeing (anxiety, depression, loss of emotional control, general positive affect and emotional ties). A single score based on all items designed as high level summary index of the person's mental health status. High scores on the Mental Health Index indicate greater psychological well being and relatively less psychological distress (range is 38-240).
Time Frame: Prior to Cycle 1 (Day -2 to +1), Every 3rd cycle (1 cycle = approx 21 days) and 6 Months Post Chemotherapy
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
Scores on a scale
  Prior to Cycle 1 | 195 [141 to 209] | 191 [165 to 230]
  Prior to Cycle 3 | 182 [120 to 228] | 189 [145 to 213]
  Prior to Cycle 6 | 196 [141 to 222] | 197 [166 to 230]
  6 Months Post Chemotherapy (+/- 15 days) | 203 [129 to 203] | 187 [179 to 233]

3. Secondary Outcome: Number of Patients With Delays In Receiving Chemotherapy Alone
Description: Number of patients who had to delay their chemotherapy treatments due to side effects.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Number; unit: participants
Arm/Group | Chemotherapy Alone
Number analyzed (Participants) | 20
participants | 8

4. Secondary Outcome: Number of Patients With Delays In Receiving Chemotherapy Plus CAM
Description: Number of patients who had to delay their chemotherapy treatments and or complementary alternative medicine due to side effects.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Number; unit: Participants
Groups:
- Chemotherapy Plus CAM: Patients receiving 6 cycles of a taxane or platinum therapy therapy for ovarian, peritoneal, or fallopian tube cancer with additional complementary alternative medicine - CAM (hypnosis, healing touch and massage therapy).
Arm/Group | Chemotherapy Plus CAM
Number analyzed (Participants) | 23
Participants | 7

5. Secondary Outcome: Average Number of Anti-Emetic Prescriptions Used After Chemotherapy Alone
Description: Determined by averaging the total number of anti-emetic prescriptions given per patient after receiving chemotherapy.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Population: Patients that received 6 cycles of chemotherapy alone.
Measure: Mean (Standard Deviation); unit: Prescriptions per participant
Arm/Group | Chemotherapy Alone
Number analyzed (Participants) | 20
Prescriptions per participant | 4.75 (0.78)

6. Secondary Outcome: Average Number of Anti-Emetic Prescriptions Used After Chemotherapy + CAM
Description: Determined by averaging the total number of anti-emetic prescriptions given per patient after chemotherapy and complementary alternative medicine.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Population: Patients receiving 6 cycles of a taxane or platinum therapy therapy for ovarian, peritoneal, or fallopian tube cancer with additional complementary alternative medicine - CAM (hypnosis, healing touch and massage therapy).
Measure: Mean (Standard Deviation); unit: Prescriptions per participant
Arm/Group | Chemotherapy Plus CAM
Number analyzed (Participants) | 23
Prescriptions per participant | 5.95 (0.81)

7. Secondary Outcome: Average Anti-Emetic Dose Use After Chemotherapy Alone
Description: Determined by averaging the total dose of anti-emetic medications given (in milligrams) per patient.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Mean (Standard Deviation); unit: Dose (mg) per participant
Arm/Group | Chemotherapy Alone
Number analyzed (Participants) | 20
Dose (mg) per participant | 453.2 (91.9)

8. Secondary Outcome: Average Anti-Emetic Dose Use After Chemotherapy Plus CAM
Description: Determined by averaging the total dose of anti-emetic medications given (in milligrams) per patient after receiving chemotherapy and complementary alternative medicine.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Mean (Standard Deviation); unit: Dose (mg) per participant
Arm/Group | Chemotherapy Plus CAM
Number analyzed (Participants) | 23
Dose (mg) per participant | 604.2 (95.5)

9. Secondary Outcome: Average Natural Killer Cell Count Levels Before Chemotherapy Alone
Description: Natural killer cells are identified as CD3 (-), CD56(+) and CD16 (+). Phenotypic analysis and measurement of NK cells (NK cell count in mm^3 drawn before chemotherapy) using flow cytometry and specific mAb.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Mean (Full Range); unit: Cells per mm^3
Arm/Group | Chemotherapy Alone
Number analyzed (Participants) | 20
Cells per mm^3 | 213 [141.3 to 257.4]

10. Secondary Outcome: Average Natural Killer Cell Count Levels Before Chemotherapy and CAM
Description: as for outcome 9
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Mean (Full Range); unit: Cells per mm^3
Arm/Group | Chemotherapy Plus CAM
Number analyzed (Participants) | 23
Cells per mm^3 | 244 [202.6 to 314.7]

11. Secondary Outcome: Comparison of Number of Patients Having Infection After Chemotherapy Alone vs. Chemotherapy Plus CAM
Description: Number of patients that had infections requiring antibiotic therapy or admission to the hospital that received either chemotherapy alone or chemotherapy plus complementary alternative medicine.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Number; unit: Participants
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
Participants | 2 | 3

12. Secondary Outcome: Comparison of Number of Patients Who Were Hospitalized After Chemotherapy Alone vs. Chemotherapy Plus CAM
Description: Count of patients who were admitted to the hospital after receiving chemotherapy treatment or chemotherapy plus complementary alternative medicine.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Number; unit: Participants
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
Participants | 5 | 6

13. Secondary Outcome: Comparison of Average White Blood Cell Count in Chemotherapy Alone vs. Chemotherapy Plus CAM
Description: Determined from white blood cell counts collected during treatment phase of study; average applied.
Time Frame: Prior to Chemotherapy through 6th Treatment with Chemotherapy (average 6 months)
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
cells/mm^3 | 5653 (695.4) | 6144 (839.3)

14. Secondary Outcome: Comparison of Average T-lymphocytes and B-lymphocytes for Chemotherapy Alone vs. Chemotherapy Plus CAM
Description: Average count determined - collected during treatment phase of study - Includes T-helper/inducer, CD4 and CD8 cells; number of CD4 and CD8 cells (in mm^3).
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
cells/mm^3
  CD4 | 680 (58.0) | 811 (82.6)
  CD8 | 281 (30.4) | 364 (34.5)

15. Secondary Outcome: Comparison of Average Salivary IgA Level in Chemotherapy Alone vs. Chemotherapy Plus CAM
Description: Determined from collection of saliva during treatment phase of study and recorded in mg/dL units.
Time Frame: Prior to Chemotherapy (Day -2 to +1) through Cycle 6 Chemotherapy (Approx. 168-180 Days)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Number analyzed (Participants) | 20 | 23
mg/dL | 14.07 (4.9) | 8.66 (1.1)

ADVERSE EVENTS:
Time Frame: From 1st Treatment through 30 Days Post Chemotherapy (approximately 7 months)
Description: Only Serious Adverse Events were collected in this study.
Arm/Group | Chemotherapy Alone | Chemotherapy + CAM
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Alone (N=20) | Chemotherapy + CAM (N=23)
Sexual/Reproductive Function (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection/Febrile Neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No